CLINICAL TRIAL: NCT03017378
Title: A Randomized, Open Clinical Trial Phase 1 Vaccine TB/FLU-01L by Intranasal and Sublingual Application for Specific Immunotherapy Pulmonary Tuberculosis
Brief Title: Reactogenicity, Safety and Immunogenicity of a TB/FLU-01L Tuberculosis Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Research Institute for Biological Safety Problems (Other Government)
Collaborators: Ministry of Health, Kazakhstan (Other Government); Research Institute of Influenza, Russia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VIT-I-01/2013
Record Dates: First submitted 2017-01-04; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Tuberculosis
Keywords: influenza vector; tuberculosis; vaccine
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TB/FLU-01L (intranasal application) (Active Comparator): Vaccine safety analysis of TB/FLU-01L at double intranasal application in healthy volunteers aged 18 to 50 years.
  Interventions: Biological: TB/FLU-01L
- TB/FLU-01L (sublingual application) (Active Comparator): Vaccine safety analysis of TB/FLU-01L at double sublingual application in healthy volunteers aged 18 to 50 years.
  Interventions: Biological: TB/FLU-01L

INTERVENTIONS:
Biological: TB/FLU-01L — TB / FLU-01L (intranasal application)
  Arms: TB/FLU-01L (intranasal application)
Biological: TB/FLU-01L — TB/FLU-01L (sublingual application)
  Arms: TB/FLU-01L (sublingual application)

SUMMARY:
The study is a single centre, phase I, open, randomized, by intranasal and sublingual application trial that explored the safety and immunogenicity of 2 doses (Day 1 and Day 21) TB/FLU-01L tuberculosis vaccine in BCG-vaccinated healthy adult subjects aged 18-50 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy BCG-vaccinated male or female adult 18 through 50 years of age at the enrollment visit.
* Literate and willing to provide written informed consent.
* A signed informed consent.
* Capable and willing to complete diary cards and willing to return for all follow-up visits.
* For females, willing to take reliable birth control measures throughout the entire period of participation in the study

Exclusion Criteria:

* Clinical, radiological (chest X-ray) or laboratory evidence of active or past TB disease.
* Current or past administration of anti-TB therapy.
* History of contact with TB patients.
* Positive QuantiFERON-TB Gold test.
* BCG vaccination in less than 6 months prior to study.
* Practice of nasal irrigation on a regular basis within the past six months or has engaged in nasal irrigation within two weeks prior to enrollment.
* Recent history of frequent nose bleeds (>5 within the past year).
* Clinically relevant abnormal paranasal anatomy.
* Recent history (within the past month) of rhino or sinus surgery, or surgery for any traumatic injury of the nose.
* Current or recent (within two weeks of enrollment) acute respiratory illness with or without fever.
* Hypersensitivity after previous administration of any vaccine.
* History of chronic alcohol abuse and/or illegal drug use.
* Any clinically significant abnormal laboratory finding.
* A positive pregnancy test for all women of childbearing potential.
* Administration of immunosuppressive drugs or other immune modifying drugs within 4 weeks prior to study enrollment.
* Acute or chronic clinically significant pulmonary disease, cardiovascular disease, gastrointestinal disease, liver disease, neurological illness, liver disease, blood disease, skin disorder, endocrine disorder, neurological illness and psychiatric disorder as determined by medical history, physical examination or clinical laboratory screening tests, which in the opinion of the investigator, might interfere with the study objectives.
* History of leukemia or any other blood or solid organ cancer.
* Seropositive for HIV, hepatitis B surface antigen and/or hepatitis C antibodies.
* Receipt of antivirals, antibiotics, immunoglobulins or other blood products within 4 weeks prior to study enrollment or planned receipt of such products during the period of subject participation in the study.
* Participation in another clinical trial within the previous three months or planned enrollment in such a trial during the period of this study.
* Subjects who are, in the opinion of the investigator, at significantly increased risk of non-cooperation with requirements of the study protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-10; Primary Completion 2014-04 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AE) - Immediate reactions | Two hours
  Commonly Solicited Local reactions associated with injections: pain, erythema/redness, swelling, induration, bruising at the injection site.
Solicited local and systemic reactions | Greater than 2 hours after administration of any dose of vaccine through 7 days following any dose
  Commonly Solicited general symptoms: fever (oral temperature ≥ 38.0°C), chills, muscle aches/myalgia, arthralgia, fatigue, malaise, headache, rash, sweating, nausea, vomiting, diarrhea and potential indicators of oculo-respiratory syndrome* (ORS).
Unsolicited AEs | Greater than 2 hours after administration of any dose of vaccine or placebo through 7 days following any dose
  Unsolicited AEs are any untoward medical occurrence in the subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Serious adverse events (SAEs), including abnormal laboratory findings | Three weeks of receipt of any dose
  Serious adverse events (SAEs) are medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.

CONTACTS AND LOCATIONS:
Overall Officials: Berik M Khairullin, PhD, Principal Investigator — Research Institute for Biological Safety Problems
Locations (1):
- National Center for Tuberculosis Problems, Kazakhstan, Almaty Qalasy, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: Undecided